CLINICAL TRIAL: NCT04673617
Title: A Multi-Center, Open-Label, Phase 1/2 Clinical Trial to Evaluate the Safety and Anti-Tumor Activity of AB-101 Monotherapy and AB-101 With Immunotherapy in Patients With Relapsed/Refractory Non-Hodgkin Lymphoma of B-Cell Origin.
Brief Title: AB-101 as Monotherapy and With Immunotherapy in Patients With Relapsed/Refractory B-Cell Non-Hodgkin Lymphoma
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Artiva Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AB-101-01
Record Dates: First submitted 2020-12-04; First posted 2020-12-17 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Non Hodgkin Lymphoma
Keywords: lymphoma; NHL; cell therapy; rituximab; NK cell; bendamustine
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma | interventions — Rituximab; Interleukin-2; Cyclophosphamide; fludarabine; Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phase 1: Dose confirmation of AB-101 as mono, ritux combo (including DLBCL specific) & BR combo (Experimental): Phase 1: Dose confirmation of AB-101 as monotherapy, in combination with rituximab (including the DLBCL specific cohort) and in combination with bendamustine and rituximab
  Interventions: Drug: AB-101; Drug: Rituximab; Drug: Interleukin-2; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Bendamustine
- Phase 2: AB-101 given with rituximab or with BR to patients with B-cell NHL at the R2PD (Experimental): Phase 2: AB-101 given with rituximab or with bendamustine and rituximab to patients with B-cell NHL at the R2PD
  Interventions: Drug: AB-101; Drug: Rituximab; Drug: Interleukin-2; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Bendamustine

INTERVENTIONS:
Drug: AB-101 — NK cell therapy
Drug: Rituximab — Anti-CD20 antibody therapy
Drug: Interleukin-2 — Immune cytokine
Drug: Cyclophosphamide — Lymphodepleting chemotherapy
Drug: Fludarabine — Lymphodepleting chemotherapy
Drug: Bendamustine — Chemoimmunotherapy

SUMMARY:
AB-101 is an off-the shelf, allogeneic cell product made of "natural killer" cells, also called NK cells. White blood cells are part of the immune system and NK cells are a type of white blood cell that are known to kill cancer cells.

This clinical trial will enroll patients with relapsed/refractory non-Hodgkin lymphoma of B-cell origin and is conducted in two phases. The primary objectives of Phase 1 are as follows: 1) to evaluate the safety of AB-101 given alone or in combination with rituximab (including the DLBCL specific cohort) or in combination with bendamustine and rituximab; 2) to evaluate the potential clinical activity of AB-101 when given in combination with rituximab or in combination with bendamustine and rituximab (combination cohorts only); and 3) to identify the recommended Phase 2 dose (RP2D). The primary objective of Phase 2 is to determine whether AB-101 in combination with rituximab or in combination with bendamustine and rituximab has anti-cancer activity in patients.

Patients will be assigned to receive either AB-101 alone as monotherapy, in combination with rituximab (including DLBCL specific cohort) or in combination with bendamustine and rituximab. All patients will receive at least 1 treatment cycle of AB-101, followed by scheduled assessments of overall health and tumor response. Patients receiving AB-101 in combination with rituximab may receive up to 3 additional cycles of treatment. Patients receiving AB-101 in combination with bendamustine and rituximab may receive up to 5 additional cycles of treatment. Patients enrolled into the DLBCL specific cohort receiving AB-101 in combination with rituximab may receive up to 3 cycles of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of aggressive NHL of B-cell origin. For enrollment into the DLBCL specific cohort: DLBCL, High-grade B-cell Lymphoma or PMBCL.
* Patient must have progressed or demonstrated intolerance to at least two lines of FDA-approved therapies, one of which must have included anti-CD20 monoclonal antibody therapy. The following are permitted: Prior autologous hematopoietic stem cell transplantation, prior treatment with FDA-approved CAR-T therapy, and/or prior treatment with an investigational agent. Prior treatment(s) with an FDA-approved CAR-T cell therapy or other cell therapies is permitted as long the patients are not considered to be refractory to this previous cell therapy approach (defined as progression within 120 days from the infusion of the cell therapy approach).
* Patient must have disease that allows for response assessment using the Lugano classification criteria.
* Ability to understand and sign the ICF.

Exclusion Criteria:

* Active CNS lymphoma or CNS involvement unless there is a history of at least 3 months of sustained remission of treated disease.
* History of clinically significant structural cardiac disease.
* Cardiac ejection fraction of < 45% on echocardiogram or MUGA scan at screening assessment.
* Inadequate pulmonary function.
* History of a solid organ allograft, or an inflammatory or autoimmune disease likely to be exacerbated by IL-2.
* Ongoing uncontrolled systemic infections.
* Positive HIV PCR test
* Positive for Hepatitis B or Hepatitis C
* Prior allogeneic stem cell transplant.
* Females of childbearing potential must be willing and able to use appropriate contraception for duration of trial and for 6 months following final AB-101 dose. Males must be sterile or commit to using appropriate contraception until 90 days following the final dose of AB-101.
* Individuals who are pregnant or lactating are ineligible.
* Patients who received a previous genetically modified cell therapy product (e.g., CD19 CAR-T), and progressed within 120 days from the time of the cell therapy infusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Safety and tolerability of AB-101 as monotherapy, and in combination with rituximab (including the DLBCL specific cohort) and in combination with bendamustine and rituximab. | From the ICF signature through 13 weeks after last study drug dose.
  Based on incidence, severity, and dose relationship of AEs and serious AEs (SAEs)
Phase 1, combination therapy: AB-101 clinical activity, determined by ORR | From baseline disease assessment through end of study participation.
  Objective response rate (ORR) is defined as the proportion of patients with a documented complete response or partial response (CR + PR) in the absence of earlier disease progression.
Phase 1, combination therapy: Identify the recommended Phase 2 dose (R2PD) for AB-101. | From ICF signature through 13 weeks after last study drug dose.
  R2PD will be determined based on safety and tolerability of AB-101 in combination with rituximab or in combination with bendamustine and rituximab.
Phase 2: Determine the efficacy profile of AB-101 in combination with rituximab or in combination with bendamustine and rituximab when administered to patients with R/R NHL of B-cell origin. | From baseline disease assessment through end of study participation.
  The efficacy profile will be determined by the ORR.

CONTACTS AND LOCATIONS:
Overall Officials: Subhashis Banerjee, M.D., Study Director — Artiva Biotherapeutics
Locations (20):
- United States (20):
  - Artiva Clinical Trial Site, Birmingham, Alabama
  - Artiva Clinical Trial Site, Tucson, Arizona
  - Artiva Clinical Trial Site, Orange, California
  - Artiva Clinical Trial Site, San Diego, California
  - Artiva Clinical Trial Site, Gainesville, Florida
  - Artiva Clinical Trial Site, Atlanta, Georgia
  - Artiva Clinical Trial Site, Chicago, Illinois
  - Artiva Clinical Trial Site, Iowa City, Iowa
  - Artiva Clinical Trial Site, Wichita, Kansas
  - Artiva Clinical Trial Site, Louisville, Kentucky
  - Artiva Clinical Trial Site, Detroit, Michigan
  - Artiva Clinical Trial Site, Lake Success, New York
  - Artiva Clinical Trial Site, New York, New York
  - Artiva Clinical Trial Site, Columbus, Ohio
  - Artiva Clinical Trial Site, Portland, Oregon
  - Artiva Clinical Trial Site, Philadelphia, Pennsylvania
  - Artiva Clinical Trial Site, Providence, Rhode Island
  - Artiva Clinical Trial Site, Dallas, Texas
  - Artiva Clinical Trial Site, Salt Lake City, Utah
  - Artiva Clinical Trial Site, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No
AlloNK is early in clinical development, next steps will be based on the progress of our data.